CLINICAL TRIAL: NCT05799092
Title: Invasive Versus Non-invasive Approach in Symptomatic Patients With Non-High Risk Coronary Artery Stenosis (SMART-STEP Trial)
Brief Title: Invasive Versus Non-invasive Approach in Symptomatic Patient With Non-High Risk Coronary Artery Stenosis
Acronym: SMART-STEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: SMC2023-02-096-001
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Computed Tomography Angiography; Non-High Risk Obstructive CAD; Diagnostic Approach; Invasive Coronary Angiography; Non-Invasive Functional Test
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Pragmatic, prospective, multi-center, open label, randomized controlled, superiority trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical outcome assessment will be performed under blinded assessment about the allocated treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive approach group (Experimental): Invasive coronary angiography will be performed as next diagnostic step in symptomatic patients with non-high risk obstructive CAD on CCTA..
  Interventions: Diagnostic Test: Invasive coronary angiography
- Non-invasive approach group (Active Comparator): Usual care of non-invasive ischemia testing (exercise electrocardiography [ECG], stress echocardiography by exercise or pharmacologic agent, nuclear test including SPECT or PET, stress cardiac magnetic resonance [MR]) will be performed as next diagnostic step in symptomatic patients with non-high risk obstructive CAD on CCTA.
  Interventions: Diagnostic Test: Non-invasive functional test

INTERVENTIONS:
Diagnostic Test: Invasive coronary angiography — As alternative to non-invasive functional testing, invasive coronary angiography will be performed.
  Arms: Invasive approach group
Diagnostic Test: Non-invasive functional test — Standard non-invasive functional testing will be performed.
  Arms: Non-invasive approach group

SUMMARY:
A pragmatic, prospective, multi-center, open label, randomized controlled, superiority trial.

The study will compare clinical outcomes between invasive versus non-invasive approach as next diagnostic step in symptomatic patients with non-high risk obstructive coronary artery disease (CAD) on coronary computed tomography-angiography (CCTA).

DETAILED DESCRIPTION:
CCTA has been emerged as useful diagnostic tool to evaluate CAD. Besides high diagnostic accuracy, CCTA has additional benefit of measuring the cumulative atherosclerotic burden and more accurately discriminating obstructive CAD with additional fractional flow reserve by CT (FFRCT), making it more predictive of a patient's prognosis. Recently, several randomized clinical trials have demonstrated the clinical utility of CCTA when compared with noninvasive stress test, which has been previously widely used as an initial assessment for stable chest pain, or invasive coronary angiography, which is the gold standard for diagnosing obstructive CAD.

On this background, CCTA, along with stress imaging test, is recommended as first step to diagnose obstructive CAD in patients with intermediate to high pretest probabilities with stable chest pain and is increasingly utilized. Although CCTA is increasingly used as initial assessment tool in these patients, there are insufficient studies to clearly establish the next step after obstructive CAD is confirmed in CCTA. Without high-risk features of CAD on CCTA, current guidelines suggest noninvasive stress imaging or FFRCT as class IIA recommendation. However, supporting evidence of these suggestions are mostly based on studies with low level of evidence. Furthermore, given the limited diagnostic performance of noninvasive stress test, concern remains whether it is safe to defer invasive coronary angiography based on the result from noninvasive stress test in patients with obstructive CAD on CCTA.

Therefore, this trial aims to compare clinical outcomes between invasive versus non-invasive approach as next diagnostic step in symptomatic patients with non-high risk obstructive CAD on CCTA.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥19 years old
2. Patients with new or worsening chest pain syndrome, equivalent symptoms, or abnormal laboratory test findings (suspected ischemic changes in electrocardiography, regional wall motion abnormality in echocardiography, or coronary calcium score > 100) suspected for clinically significant CAD who are evaluated by CCTA
3. Any other clinical circumstance in which physician judged to proceed CCTA
4. Obstructive CAD in CCTA (≥50% diameter stenosis)
5. Subject who can verbally confirm understandings of risks, benefits, and treatment alternatives of receiving invasive approach and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria:

1. Diagnosed or suspected acute coronary syndrome (ACS) requiring hospitalization or urgent or emergent testing (elevated cardiac troponin or CK-MB)
2. High risk CAD (left main stenosis ≥ 50%; anatomically significant 3-vessel disease with ≥70% stenosis)
3. Hemodynamically or clinically unstable condition (systolic BP < 90 mmHg, ventricular arrhythmias, or persistent resting chest pain in ischemic nature despite adequate therapy
4. Known CAD with previous MI, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG)
5. Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
6. Known significant congenital, severe valvular or cardiomyopathic (hypertrophic or dilated cardiomyopathy, or any other forms) process which could explain cardiac symptoms.
7. Severe left ventricular systolic dysfunction (ejection fraction <30%)
8. Intolerance to Aspirin, Clopidogrel, or Heparin.
9. Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment)
10. Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first event of major adverse cardiac events (MACE) | 2 years after the last patient enrollment
  MACE is a composite of death from any causes, myocardial infarction (MI), clinically driven unplanned revascularization.

SECONDARY OUTCOMES:
All-cause death | 2 years after the last patient enrollment
  All-cause death
Cardiac death | 2 years after the last patient enrollment
  Cardiac death
Any MI | 2 years after the last patient enrollment
  Defined by Forth Universal definition of MI
Spontaneous MI | 2 years after the last patient enrollment
  Defined by Forth Universal definition of MI
Procedure-related MI | 2 years after the last patient enrollment
  Defined by ARC II definition
Resuscitated cardiac arrest | 2 years after the last patient enrollment
  Resuscitated cardiac arrest
Unplanned revascularization (clinically driven) | 2 years after the last patient enrollment
  Unplanned revascularization (clinically driven)
Cerebrovascular accidents | 2 years after the last patient enrollment
  Cerebrovascular accidents (ischemic or hemorrhagic)
Major adverse cardiac and cerebrovascular events | 2 years after the last patient enrollment
  Major adverse cardiac and cerebrovascular events (MACCE, a composite of death, MI, clinically-driven unplanned revascularization, or cerebrovascular accident)
Rate of index coronary angiography | up to 30 days following randomization
  Rate of index coronary angiography
Rate of index revascularization by PCI or CABG | up to 30 days following randomization
  Rate of index revascularization by PCI or CABG
European Quality of Life-5 Dimensions | 6 months after initial management according to allocated diagnostic test
  European Quality of Life-5 Dimensions
Seattle Angina Questionnaire | 6 months after initial management according to allocated diagnostic test
  Seattle Angina Questionnaire
Total medical cost | 2 years after the last patient enrollment
  Total medical cost
Procedure-related complications from invasive procedure | up to 30 days following randomization
  Procedure-related complications from invasive procedure

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (22):
- South Korea (22):
  - SoonChunHyang University Hospital Bucheon, Bucheon-si
  - Kangwon National University Hospital, Chuncheon
  - Chungbuk National University Hospital, Chungju
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Inje university Ilsan Paik hospital, Ilsan
  - Gachon University Gil Medical Center, Incheon
  - Kwandong University Intl. ST. Mary's Hospital, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Hanyang University Seoul Hospital, College of Medicine, Hanyang University, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Access Criteria: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked